CLINICAL TRIAL: NCT01920204
Title: Phase II Single Arm Open Pilot Study to Demonstrate the Efficacy of Midostaurin in Symptom Improvement and Decrease of Mast Cell Burden in Patients With Indolent or Smoldering Systemic Mastocytosis.
Brief Title: Midostaurin in Indolent Systemic Mastocytosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Prof.dr. J.C. Kluin-Nelemans, Prof.dr., University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCG41973
Record Dates: First submitted 2013-08-07; First posted 2013-08-09 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Indolent Systemic Mastocytosis
Keywords: Mastocytosis; ISM; SSM
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis | interventions — midostaurin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Midostaurin (Experimental): Treatment with Midostaurin, twice daily 100 mg orally for 6 months continuously.
  Interventions: Drug: Midostaurin,

INTERVENTIONS:
Drug: Midostaurin, — Midostaurin, twice daily 100 mg orally, continuously for 6 months
  Other Names: PKC412

SUMMARY:
Rationale: Patients with indolent or smoldering systemic mastocytosis can have severe disabling symptoms. Almost all patients have fatigue, a compromised quality of life, hampering normal functioning. Because this form of mastocytosis is not considered life-threatening, mast cell eradication has never been applied and patients receive only symptomatic therapy with histamine blockers. Midostaurin, a c-KIT inhibitor has shown activity regarding symptom control and decrease of malignant mast cells in patients with aggressive systemic mastocytosis (ASM) or mast cell leukemia

DETAILED DESCRIPTION:
Objective:

Primary: To study in a pilot phase II trial the efficacy of midostaurin administered at an oral dose of 100 mg twice daily in patients with indolent or smoldering systemic mastocytosis on mediator symptom reduction, documented by the Mastocytosis Symptom Assessment Questionnaire, measured at 3 months.

Secondary:

1. To study whether symptom improvement persists at 6 months, and whether midostaurin can reduce mast cell infiltration in the skin and bone marrow, documented by decrease of serum tryptase, decrease of urticaria pigmentosa and decrease of bone marrow mast cells.
2. To assess safety and tolerability of midostaurin in the above mentioned settings

Study design: Single arm, open label pilot phase II study.

Study population: Adult patients (n=20) with histologically documented systemic mastocytosis, indolent or smoldering subtype, with severe symptoms, not controlled by histamine 1 and 2 blockers.

Intervention: treatment with Midostaurin, twice daily 100 mg orally for 6 months continuously.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Indolent Systemic Mastocytosis (ISM) or Smouldering Systemic Mastocytosis (SSM) according to the WHO criteria
* Presence of the D816V c-KIT mutation
* Serum tryptase > 20 mg/l
* Serious mediator-related symptoms that cannot be controlled by H1 and H2 blocking drugs. Symptoms will be scored by an adapted MSAF (mastocytosis symptom assessment form) with at least:

  * a pre-study score of 4 or more on 3 non-related items,
  * or a pre-study score of 5 or more on 2 non-related items.
  * one item from the scoring list can be replaced by flushes 7 or more per week or anaphylactic attacks 1 or more per week.
* Age >18 years
* Willingness to apply optimal contraceptive measures (double barrier method, both men and women) for women below the age of 55, men at all ages; for both: if sexually active.
* Written informed consent

Exclusion Criteria:

* Aggressive systemic mastocytosis, mast cell leukemia, or ASM with or without accompanying non-clonal related non-mast cell disorder (SM-ANHMD).
* Any known other present malignancy, non-melanoma skin cancers excluded
* History of malignancy within the last 5 years, non-melanoma skin cancers excluded
* Any serious comorbidity interfering with therapy compliance and follow-up compliance
* Pregnancy
* Patients not willing or who are not able to comply with contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-03 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Symptom Scoring | 12 weeks
  Percent change in the total score ("Sumscore") of all symptoms assessed by the Mastocytosis Symptom Assessment Form (MSAF) after 12 weeks.

SECONDARY OUTCOMES:
Persistence of improvements | 6 months
  persistence of improvement symptom score at 6 months.
Mast cell burden | 6 months
  Percent change in the mast cell burden (bone marrow infiltrate, skin infiltrate, serum tryptase levels) after 6 months.
Adverse events | 6 months
  Number and grading of Common Terminology Criteria adverse events during the 6 months of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: J.C. Kluin-Nelemans, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Derived] van Anrooij B, Oude Elberink JNG, Span LFR, de Monchy JGR, Rosati S, Mulder AB, Kluin-Nelemans JC. Midostaurin in patients with indolent systemic mastocytosis: An open-label phase 2 trial. J Allergy Clin Immunol. 2018 Sep;142(3):1006-1008.e7. doi: 10.1016/j.jaci.2018.06.003. Epub 2018 Jun 8. No abstract available. PMID 29890238